CLINICAL TRIAL: NCT00097123
Title: RCT of Misoprostol for Postpartum Hemorrhage in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Missouri-Columbia (Other); Jawaharlal Nehru Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GN 08; U01HD042372 (NIH)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Postpartum Hemorrhage; Pregnancy
Keywords: Acute postpartum hemorrhage; PPH; Misoprostol; Global Network; Uterotonics; India; Maternal and child health; International; Women's health
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
Death rates for pregnant women in rural India are approximately forty-five times higher than in the United States. Bleeding after the birth of a child and underlying anemia are the primary causes of mothers' deaths and sickness in rural India. This study assesses the effectiveness of an oral drug, misoprostol, given in the late stage of labor to reduce the incidence of maternal bleeding following births assisted by midwives in selected sites in Belgaum District, Karnataka, India.

DETAILED DESCRIPTION:
Despite existing knowledge of ways to effectively treat postpartum hemorrhage (PPH), lack of resources in rural India has impeded improvement in rates of maternal mortality and morbidity. Most births take place at home, and local auxiliary nurse midwives are not trained or certified to administer injectable uterotonics. Reduction in postpartum hemorrhage may decrease other adverse maternal outcomes such as the need for additional uterotonic agents, blood transfusion, surgical intervention or death. The main hypothesis of the study is that misoprostol administered orally during the third stage of labor will significantly reduce the incidence of acute postpartum hemorrhage. The advantages of misoprostol are: that it is relatively inexpensive, is an oral preparation of 600 mcg with a long shelf life, and does not require refrigeration. One thousand six hundred women giving birth in selected sites in Belgaum District, Karnataka, India will be randomly assigned to misoprostol or placebo. The primary outcome is the incidence of acute postpartum hemorrhage; secondary outcomes include incidence of delayed postpartum hemorrhage and secondary infection; transport to higher-level facility; use of uterotonic agents; blood transfusion; and maternal mortality for 42 days. A nested case-control analysis of women who experience acute severe postpartum hemorrhage, compared to women who do not, will identify socioeconomic, behavioral, cultural, and systems factors associated with postpartum hemorrhage. For purposes of this study, acute PPH is defined as blood loss equal to or greater than 500 ml within 2 hours of delivery and acute severe PPH as blood loss equal to or greater than 1000 ml within 2 hours of delivery.

The sample size was based on a decrease of 50% PPH in the treated versus the control group; 20% rate of non-compliance, power of 96%, and a two-tailed type I error of 0.05

ELIGIBILITY:
Inclusion Criteria:

* Gestational age equal to or greater than 28 weeks pregnant
* Planning to deliver at home or at a sub-center in the Belgaum District, Karnataka India
* Anticipating a spontaneous vaginal delivery
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Previous caesarian section
* Scheduled for caesarian section
* Hemoglobin level less than 8 Gms%
* Episodes of antepartum bleeding during the current pregnancy
* Blood pressure more than 140 mm of Hg systolic and 90 mm of Hg diastolic
* In active labor and not previously screened, recruited, and consented
* Absence of fetal heart sounds
* Multiple pregnancy
* Known history of bronchial asthma
* Prior enrollment in this study during a previous pregnancy
* History of complications (ante/postpartum hemorrhage/retained placenta/ acute inversion of uterus) during a previous pregnancy
* High risk conditions including: diabetes, cardiac ailments, seizures, placenta previa or anticipated breech delivery.
* Receiving injectable medicine at time of delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2002-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Incidence of acute postpartum hemorrhage: blood loss ≥ 500 ml within two hours of delivery

SECONDARY OUTCOMES:
Incidence of delayed postpartum hemorrhage and secondary infection (lower abdominal pain, fever and foul discharge)
Transport to higher-level medical facility
Use of uterotonic agents
Blood transfusion
Surgical intervention including curettage, vacuum aspiration for retained placental tissue or hysterectomy
Maternal mortality for 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Derman, M.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- KLE Society's Jawaharlal Nehru Medical College, Belagavi, Karnataka, India

REFERENCES:
- [Result] Derman RJ, Kodkany BS, Goudar SS, Geller SE, Naik VA, Bellad MB, Patted SS, Patel A, Edlavitch SA, Hartwell T, Chakraborty H, Moss N. Oral misoprostol in preventing postpartum haemorrhage in resource-poor communities: a randomised controlled trial. Lancet. 2006 Oct 7;368(9543):1248-53. doi: 10.1016/S0140-6736(06)69522-6. PMID 17027730
- See also: Website for the Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org